CLINICAL TRIAL: NCT04913324
Title: The RECOVER Study - Remote Early Intervention for Cerebral Palsy to Improve Outcomes Using Virtual Care Following pERinatal Asphyxia
Brief Title: Early Virtual Intervention for Infants With CP Following HIE Diagnosis
Acronym: RECOVER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Linh Ly, Medical Director, NICU and Neonatal Neurodevelopmental Follow-up Clinic, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1000064940
Record Dates: First submitted 2021-04-07; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Cerebral Palsy; Hypoxic-Ischemic Encephalopathy; Brain Injuries; Perinatal Hypoxia
Keywords: HIE; Cerebral Palsy; Infant; Virtual Care; Hypoxic-Ischemic Encephalopathy; Follow-Up; Brain Injuries; Perinatal Hypoxia
MeSH Terms: conditions — Cerebral Palsy; Hypoxia-Ischemia, Brain; Brain Injuries | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: 18 month follow-up assessment will be completed by a blinded clinician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Care (Experimental)
  Interventions: Behavioral: Virtual Care
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Virtual Care — Infants randomized at 4 months of age to the intervention arm will participate in virtual care visits for 16 weeks in addition to standard of care in-hospital visits.
  Arms: Virtual Care

SUMMARY:
This will be a five year study that will be a prospective, randomized, controlled trial (RCT) to assess the effect of a virtual early intervention care delivery model in the provision of therapy to enhance the neurodevelopmental trajectory of infants with brain injury. In addition, the investigators will enhance understanding of the social and parental contributors to outcomes and the early health economic impact of a virtual clinic. The results of this study will help inform the design of a larger, multi-center randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of moderate to severe hypoxic ischemic encephalopathy as defined based on Sarnat criteria 35
2. Received therapeutic hypothermia
3. Abnormal brain MRI (deep grey matter, watershed or mixed patterns of injury) in the first seven days of life
4. Greater than or equal to 34 weeks gestation
5. Patients are followed by the Neonatal Follow-Up Clinic at SickKids
6. Abnormal GMA (abnormal or absent fidgety movements) at 12 weeks of age

Exclusion Criteria:

1. Known or high suspicion of a genetic syndrome
2. Residence post-discharge will not be with biological parents
3. Limited fluency in English
4. No internet access

Ages: 4 Months to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor outcomes at 18 months between groups using the the motor function score as measured using the Bayley Scales of Infant and Toddler Development | 18 months

SECONDARY OUTCOMES:
Correlation between parent mental health using the modified Perinatal PTSD Questionnaire, Parent Stress Index, and neurodevelopmental outcomes of patients at 18 months using the Bayley Scales of Infant and Toddler Development | 18 months
Sociodemographic factors that contribute to improved neurodevelopmental outcomes at 18 months as reported using a Sociodemographics Questionnaire | 18 months
Cost-effectiveness of providing remote, early, intensive therapy for children at risk for cerebral palsy versus standard of care as reported using a Health Economics Questionnaire. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Linh Ly, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Kalaf H, Martinez A, Danguecan A, Christensen R, Tam EWY, Chau V, Wilson D, Tung S, Branson HM, Ly LG, Cizmeci MN. The Prognostic Weight of Clinical, Biochemical, Electrographic, and Neuroimaging Biomarkers in Perinatal Hypoxic-Ischemic Encephalopathy Spectrum. J Pediatr. 2025 Oct 31;289:114885. doi: 10.1016/j.jpeds.2025.114885. Online ahead of print. PMID 41177395
- [Derived] Raghu K, Kalish BT, Tam EWY, El Shahed A, Chau V, Wilson D, Tung S, Kazazian V, Miran AA, Hahn C, Branson HM, Ly LG, Cizmeci MN. Prognostic Indicators of Reorientation of Care in Perinatal Hypoxic-Ischemic Encephalopathy Spectrum. J Pediatr. 2025 Jan;276:114273. doi: 10.1016/j.jpeds.2024.114273. Epub 2024 Aug 30. PMID 39216619